CLINICAL TRIAL: NCT01060501
Title: Phase 3 Study of Adjuvant Chemoradiotherapy of Advanced Resectable Rectal Cancer Comparing Modulation of 5-FU With Folinic Acid or With Interferon-alpha
Brief Title: Modulation of Adjuvant 5-FU by Folinic Acid and Interferon-alpha in Colon Cancer
Acronym: FOGT1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Medac GmbH (Hamburg, Germany) (Unknown); Roche (Grenzach-Wyhlen, Germany) (Unknown)
Responsible Party: Prof. Dr. Marko Kornmann, Study Group Oncology of Gastrointestinal Tumors (FOGT)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOGT1
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 1991-07

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; adjuvant chemoradiotherapy; 5-FU, interferon-alpha; Locally advanced resectable rectal cancer (UICC stage II and III)
MeSH Terms: conditions — Rectal Neoplasms | interventions — Leucovorin; Interferon-alpha

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 5-FU (Active Comparator): Standard arm Systemic drug administration of 5-FU (intravenous)
  Interventions: Drug: Folinic Acid, interferon-alpha
- 5-FU + folinic acid (Experimental): Experimental arm Systemic drug administration of 5-FU + folinic acid (intravenous)
  Interventions: Drug: Folinic Acid, interferon-alpha
- 5-FU + Interferon-alpha (Experimental): Experimental arm Systemic drug administration of 5-FU + interferon-alpha (intravenous)
  Interventions: Drug: Folinic Acid, interferon-alpha

INTERVENTIONS:
Drug: Folinic Acid, interferon-alpha — 5-FU, 450 mg/m² i.v. for 60 min, weekly for 52 weeks postoperatively Folinic acid, 200 mg/m² i.v. 10 min, weekly for 52 weeks postoperatively 6x10 (high6) I.U. as subcutaneous self injection 3x weekly. Training of self injection was initiated on day 28 (duration until week 52)

SUMMARY:
The primary objective was to improve adjuvant 5-FU chemoradiotherapy in resectable rectal cancer. The investigators hypothesis was that modulation of 5-FU by addition of either FA or INF-alpha may increase overall survival.

DETAILED DESCRIPTION:
Primary endpoint was overall survival (OS). For sample size estimation the following assumptions were made: The 5-year OS rate of 5-FU was estimated to be 58%. Our intention was to detect an increase in the 5-year OS rate by one of the additives of at least 10% with a power of 80% and a level of significance of 5% in comparison to 5-FU (one-sided). Hypotheses were analyzed as pair wise comparisons between the treatment options. This resulted in a target sample size of 280 patients per group and a total of 840 patients.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility was defined as potentially curative en-bloc resection (R0) of an adenocarcinoma of the rectum with a lower tumor edge within 12 cm from the anal verge determined by rectoscopy, a pathologic UICC stage II (pT3/4pN0M0) or III (pT1-4pNposM0) with examination of at least 12 lymph nodes, a white blood count ≥ 3,500/µl, a platelet count ≥ 100,000/µl, a ECOG performance status of 0 or 1, and written informed consent.

Exclusion Criteria:

* Ineligible were patients not fulfilling these criteria or having a history of cancer except for adequately treated superficial basal or squamous cell skin cancer or in situ carcinoma of the cervix, getting previous radio- or chemotherapy, pregnant or nursing women, other having severe concomitant diseases limiting life expectancy or not allowing chemotherapy, and with social conditions not allowing a 5-year follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 1992-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
overall survival | 5-year

SECONDARY OUTCOMES:
recurrence-free survival | 5-year
Toxicity (WHO) | 5-year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General, Visceral, and Transplantation Surgery, University of Ulm, Ulm, Germany